CLINICAL TRIAL: NCT05364554
Title: A Phase 2b Multicenter, Long-Term Extension, Dose-ranging Study to Evaluate the Efficacy and Safety of JNJ-77242113 for the Treatment of Moderate-to-Severe Plaque Psoriasis
Brief Title: A Long-term Extension Study of JNJ-77242113 in Participants With Moderate-to-Severe Plaque Psoriasis
Acronym: FRONTIER 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109155; 2021-004320-16 (EudraCT Number); 77242113PSO2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: JNJ-77242113 Dose 1 Once Daily (QD) (Experimental): Participants originally randomized to JNJ-77242113 Dose 1 QD in originating study 77242113PSO2001 will continue to receive JNJ-77242113 Dose 1 QD from Week 0 through Week 36 in this study.
  Interventions: Drug: JNJ-77242113
- Group 2: JNJ-77242113 Dose 2 QD (Experimental): Participants originally randomized to JNJ-77242113 Dose 2 QD in originating study 77242113PSO2001 will continue to receive JNJ-77242113 Dose 2 QD from Week 0 through Week 36 in this study.
  Interventions: Drug: JNJ-77242113
- Group 3: JNJ-77242113 Dose 3 QD (Experimental): Participants originally randomized to JNJ-77242113 Dose 3 QD in originating study 77242113PSO2001 will continue to receive JNJ-77242113 Dose 3 QD from Week 0 through Week 36 in this study.
  Interventions: Drug: JNJ-77242113
- Group 4: JNJ-77242113 Dose 1 Twice Daily (BID) (Experimental): Participants originally randomized to JNJ-77242113 Dose 1 BID in originating study 77242113PSO2001 will continue to receive JNJ-77242113 Dose 1 BID from Week 0 through Week 36 in this study.
  Interventions: Drug: JNJ-77242113
- Group 5: JNJ-77242113 Dose 3 BID (Experimental): Participants originally randomized to JNJ-77242113 Dose 3 BID in originating study 77242113PSO2001 will continue to receive JNJ-77242113 Dose 3 BID from Week 0 through Week 36 in this study.
  Interventions: Drug: JNJ-77242113
- Group 6: JNJ-77242113 Dose 3 QD (Experimental): Participants originally randomized to placebo in originating Study 77242113PSO2001 will receive JNJ-77242113 Dose 3 QD from Week 0 through Week 36 in this study.
  Interventions: Drug: JNJ-77242113

INTERVENTIONS:
Drug: JNJ-77242113 — JNJ-77242113 tablet will be administered orally.

SUMMARY:
The purpose of this study is to evaluate long-term clinical response of JNJ-77242113 treatment in participants with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
The populations of people living with moderate to severe psoriasis is approximately 3.5 billion which are mostly managed with topical and conventional therapies. JNJ-77242113, investigational drug, targets the immune responses in the body and skin which impacts diseases, such as psoriasis and this study evaluates JNJ-77242113 as options of advanced therapies in moderate to severe plaque psoriasis. This is a long-term extension study of JNJ-77242113 in eligible participants who have completed the Week 16 visit of the originating Study 77242113PSO2001. The total duration of this study will be up to 40 weeks which will include a 36-week treatment period, and a 4-week safety follow-up period after the last study intervention administration. Safety will be assessed by adverse events (AEs), clinical safety laboratory assessments, electrocardiograms (ECGs), vital signs and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed the Week 16 visit in Protocol 77242113PSO2001
* In the opinion of the investigator, may benefit from inclusion in this long term extension (LTE) study
* Must agree to avoid prolonged sun exposure and avoid use of tanning booths or other ultraviolet light sources during the study
* Must agree to discontinue all topical therapies that could affect psoriasis or the psoriasis area severity index (PASI) or investigator's global assessment (IGA) evaluation, other than nonmedicated emollient and salicylic acid shampoos, prior to first administration of study intervention
* Agree not to receive a live virus or live bacterial vaccination during the study, or within 4 weeks after the last administration of study intervention

Exclusion Criteria:

* Was permanently discontinued from study intervention in Protocol 77242113PSO2001 for any reason
* Has received any biologic therapy or experimental therapy since completion of the originating study, 77242113PSO2001
* Has received any live virus or bacterial vaccination within 12 weeks before the first administration of study intervention
* Has received the bacille Calmette-Guerin (BCG) vaccine within 12 months of the first administration of study intervention
* Currently has hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or has other clinically active liver disease, or tests positive for HBsAg or anti-HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 75 Score at Week 36 | Week 36
  Percentage of participants achieving PASI 75 score (greater than or equal to [>=] 75 percent [%] improvement in PASI from baseline of the originating study [77242113PSO2001]) at Week 36 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.

SECONDARY OUTCOMES:
Percentage of Participants Achieving PASI 90 Score at Week 36 | Week 36
  Percentage of participants achieving PASI 90 score (>=90% improvement in PASI from baseline of the originating study [77242113PSO2001]) at Week 36 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Participants Achieving PASI 100 Score at Week 36 | Week 36
  Percentage of participants achieving PASI 100 score (>=100% improvement in PASI from baseline of the originating study [77242113PSO2001]) at Week 36 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Change From Baseline in PASI Total Score at Week 36 | Baseline and Week 36
  Change from baseline of the originating study (77242113PSO2001) in PASI total score at Week 36 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Participants Achieving an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) at Week 36 | Week 36
  Percentage of participants who achieve an IGA score of cleared (0) or minimal (1) at Week 36 will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Change from Baseline in Psoriasis Symptoms and Signs Diary (PSSD) Symptoms Scores at Week 36 | Baseline and Week 36
  Change from baseline of originating Study (77242113PSO2001) in PSSD symptoms scores at Week 36 will be reported. The PSSD includes patient-reported outcome (PRO) questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Change from Baseline in PSSD Signs Score at Week 36 | Baseline and Week 36
  Change from baseline of originating study (77242113PSO2001) in PSSD signs score at Week 36 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Percentage of Participants Achieving PSSD Symptoms Score=0 at Week 36 Among Participants With a Baseline (in the Originating Study) Symptoms Score >=1 | Week 36
  Percentage of participants achieving PSSD symptoms score=0 at Week 36 among participants with a baseline (in the originating study 77242113PSO2001) symptoms score >=1 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Percentage of Participants Achieving PSSD Signs Score=0 at Week 36 Among Participants With a Baseline (in the Originating Study) Signs Score >=1 | Week 36
  Percentage of participants achieving PSSD signs score=0 at week 36 among participants with a baseline (in the originating study) signs score >=1 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Number of Participants with Adverse Events (AEs) | Up to Week 40
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Number of Participants with Serious Adverse Events (SAEs) | Up to Week 40
  SAE is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (60):
- United States (14):
  - Pacific Skin Institute, Sacramento, California
  - Renstar Medical Research, Ocala, Florida
  - Forcare Clinical Research Inc, Tampa, Florida
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Indiana Clinical Trial Center, Plainfield, Indiana
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Vivida Dermatology, Las Vegas, Nevada
  - Windsor Dermatology, PC, East Windsor, New Jersey
  - Oregon Dermatology and Research Center, Portland, Oregon
  - University of Pittsburgh Department of Dermatology, Pittsburgh, Pennsylvania
  - Modern Research Associates, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Center for Clinical Studies, Webster, Texas
  - Premier Clinical Research, Spokane, Washington
- Canada (4):
  - Dermatrials Research, Hamilton, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
- France (3):
  - Centre Hospitalier Le Mans, Le Mans
  - Hopital Charles Nicolle, Rouen
  - HIA Sainte Anne, Toulon
- Germany (12):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - CRS Clinical Research Services Berlin GmbH, Berlin
  - Niesmann & Othlinghaus GbR, Bochum
  - Rosenpark Research GmbH, Darmstadt
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - Derma-Study-Center Friedrichshafen GmbH, Friedrichshafen
  - MensingDerma research GmbH, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Schleswig Holstein Kiel, Kiel
  - Gemeinschaftspraxis Scholz/Sebastian/Schilling, Mahlow
  - Hautarztpraxis, Witten
- Japan (7):
  - Takagi Dermatological Clinic, Obihiro-shi
  - Kume Clinic, Sakai
  - Sapporo Skin Clinic, Sapporo
  - Shizuoka General Hospital, Shizuoka
  - Shirasaki Dermatology Clinic, Takaoka
  - Toyama Prefectural Central Hospital, Toyama
  - Nomura Dermatology Clinic, Yokohama
- Poland (5):
  - Nzoz Zdrowie Osteo-Medic, Bialystok
  - Dermed Centrum Medyczne Sp z o o, Lodz
  - Dermodent Centrum Medyczne Aldona Czajkowska Rafal Czajkowski S C, Osielsko
  - Klinika Ambroziak Estederm Sp. z o.o, Warsaw
  - Wro Medica, Wroclaw
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - KyungHee University Hospital, Seoul
- Spain (4):
  - Hosp. Univ. Germans Trias I Pujol, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. de Manises, Valencia
- Taiwan (4):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang-Gung Memorial Hospital, LinKou Branch, Taoyuan District
- United Kingdom (2):
  - Guys and St Thomas NHS Foundation Trust, London
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Strawn D, Krueger JG, Bissonnette R, Eyerich K, Ferris LK, Paller AS, Pinter A, Richards D, Chen EY, Paget K, Horowitz D, Parast R, Rusbuldt JJ, Sendecki J, Bhagat S, Tomsho LP, Chou CH, Polak ME, Keyes BE, Bozenhardt E, Xiong Y, Zhou W, DeKlotz C, Newbold P, Waterworth DM, Miller M, Ota T, Yang YW, Leung MW, Miller LS, Cuff CA, McRae B, Ruane D, Kannan AK. Icotrokinra induces early and sustained pharmacodynamic responses in phase IIb study of patients with moderate-to-severe psoriasis. JCI Insight. 2025 Dec 22;10(24):e193563. doi: 10.1172/jci.insight.193563. eCollection 2025 Dec 22. PMID 41424381
- [Derived] LaRoche JK, Lanier J, Alvarenga R, Collins M, Costelloe T, Chiau A, Whetherly H, De Soete W, Faludi J, Rens K. Climate footprint of industry-sponsored in-human clinical trials: life cycle assessments of clinical trials spanning multiple phases and disease areas. BMJ Open. 2025 Feb 19;15(2):e085364. doi: 10.1136/bmjopen-2024-085364. PMID 39971605